CLINICAL TRIAL: NCT03826836
Title: Effectiveness of Mindfulness-based Stress Reduction for Improving Quality of Life in Patients With Cardiovascular Disease: a Randomised Controlled Trial
Brief Title: Mind Our Heart Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Dutch Heart Foundation (Other); Erasmus Medical Center (Other); Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Joep Teijink, Principal Investigator, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CZE-2018.24
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Peripheral Arterial Disease; Heart Failure; Myocardial Infarction; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Heart Failure; Myocardial Infarction; Atherosclerosis | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Treatment as usual (i.e. best medical treatment).
- Mindfulness-based stress reduction (Experimental): Treatment as usual (i.e. best medical treatment) in combination with an eight-week mindfulness-based stress reduction programme.
  Interventions: Behavioral: Mindfulness-based stress reduction

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction — Mindfulness-based stress reduction (MBSR) is a structured programme of 8 weekly sessions of 2-2,5 hours in groups of 8-16 participants organized at the hospital sites. Additionally, participants are encouraged to practice each day for 30-45 minutes using audio-recordings of the guided exercises. The programme is provided by experienced mindfulness teachers according to the standard MBSR protocol, except for the all-day session.
  Arms: Mindfulness-based stress reduction

SUMMARY:
Patients with atherosclerotic cardiovascular disease (i.e. peripheral artery disease, ischemic heart failure, myocardial infarction) are randomised to (1) treatment as usual (i.e. best medical care) or (2) treatment as usual (i.e. best medical care) in combination with an eight-week mindfulness-based stress reduction programme.

DETAILED DESCRIPTION:
Rationale: Distress, including depression, anxiety, and chronic stress, is common among patients with cardiovascular disease. This reduces their quality of life and worsens their prognosis. A structured mindfulness training programme, such as the 8-week mindfulness-based stress reduction (MBSR) course, may reduce distress, improve quality of life, support a healthy lifestyle and modify cardiovascular risks. The aim of this randomised controlled trial is to determine whether MBSR improves the quality of life in patients with atherosclerotic cardiovascular disease.

Objective: The primary objective is the effect of MBSR on quality of life. Secondary objectives are the effects of MBSR on mental health, mindfulness, and cardiovascular risk factors, and the cost-effectiveness of MBSR.

Study design: Multicenter Torgerson preference randomised controlled trial. Complemented with qualitative research in a maximum of 12 patients in the intervention arm.

Study population: Patients with atherosclerotic cardiovascular disease (i.e. coronary artery disease, ischemic heart failure, and peripheral artery disease).

Intervention: The intervention group will receive an 8-week MBSR programme in addition to treatment as usual (TAU+MBSR), while the control group will receive only treatment as usual (TAU).

Main study parameters: The primary outcome is the change of scores on the SF-36 scale, which is an instrument for measuring quality of life. Secondary outcomes are depression and anxiety (HADS questionnaire), stress (PSS-10 questionnaire), mindfulness (FFMQ-SF questionnaire), smoking, BMI, blood pressure, heart rate, plasma lipids and HbA1c, hair cortisol, quality of life measured by EQ-5D-5L questionnaire, health care costs, and non-health care costs.

Nature and extent of the burden and risks: Participation in this trial is not associated with additional risks compared to treatment as usual. MBSR is proven to be safe and is widely accepted for patients with a variety of conditions as well as for healthy persons. The burden of participation (i.e. time investment and extra examinations) will be compensated by the possible benefits. MBSR is already successfully used for the treatment of a variety of physical and mental conditions, including chronic pain, cancer, anxiety, depression and burnout. As a substantial number of patients with cardiovascular disease experience distress, mindfulness could be an effective intervention for this population as well. The American Heart Association recently stated that meditation, as it is a low-cost and low-risk intervention, may be considered as an adjunct to current cardiovascular management. However, further research on the effects of mindfulness is warranted and should preferably consist of randomised, adequately powered studies with use of a control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult (i.e. older than 18 years)
* Established ASCVD (i.e. coronary artery disease, ischemic heart failure, or peripheral artery disease)

Exclusion Criteria:

1. Current acute cardiovascular event (myocardial infarction, major stroke, acute limb ischemia in prior 2 weeks)
2. Critical limb ischemia
3. Terminal illness
4. History of psychosis
5. Current severe psychiatric disorder
6. Current psychotherapy
7. Non-Dutch speaking
8. Cognitive impairment
9. Behavioural problems that distort group therapy
10. Active mindfulness/meditation or yoga practice within the past year
11. Current participation in another clinical trial that interferes with this study's intervention or primary outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Health Related Quality of Life | Baseline, 3, 6, 12, 24, and 60 months.
  Health related quality of life (HRQOL) will be measured with the SF-36 (Short Form) questionnaire, which contains 36 questions. The total score is based on a 100-point scale, with a higher score indicating a higher quality of life.
  Physical health summary scores are derived using four scales (physical functioning, role functioning due to physical problems, bodily pain and general health perceptions), while mental health summary scores are derived using four other scales (mental health, role limitations due to emotional problems, social functioning and vitality).
  The change of scores over time for all time points will be reported.

SECONDARY OUTCOMES:
Depression | Baseline, 3, 6, 12, 24, and 60 months.
  Depression will be measured with the Hospital Anxiety and Depression Scale (HADS), which is a 14-item self-report screening scale which is used to indicate the possible presence of anxiety and/or depressive symptoms. The scale includes 7 items on anxiety and 7 items on depression, both with a score ranging from 0 to 21. The total score is classified into no anxiety or depression disorder (≤7), possible disorder (8-10), and probable disorder (≥11).
Anxiety | Baseline, 3, 6, 12, 24, and 60 months.
  Anxiety will be measured with the Hospital Anxiety and Depression Scale (HADS), which is a 14-item self-report screening scale which is used to indicate the possible presence of anxiety and/or depressive symptoms. The scale includes 7 items on anxiety and 7 items on depression, both with a score ranging from 0 to 21. The total score is classified into no anxiety or depression disorder (≤7), possible disorder (8-10), and probable disorder (≥11).
Perception of stress | Baseline, 3, 6, 12, 24, and 60 months.
  Stress will be measured with the Perceived Stress Scale 10, which is the most widely used psychological instrument for measuring the perception of stress and consists of 10 items. It is a measure of the degree to which situations in one's life are appraised as stressful. Items are designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. Scores can range from 0 to 40 with higher scores indicating higher perceived stress.
Hair cortisol levels | Baseline, 3, 6 and 12 months.
  Measurement of cortisol levels in hair
Five facets of mindfulness | Baseline, 3, 6, 12, 24, and 60 months.
  Mindfulness will be measured with the Five Facet Mindfulness Questionnaire Short-Form (FFMQ-SF), and a single question about daily mindfulness practice (daily, weekly or not regularly).
  The FFMQ-SF is a 24-items self-report screening scale which is used to measure five facets of mindfulness. These five facets are observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Facet scores range from 5 to 25 (for the 'observing' facet 4 to 20), with higher scores indicating more mindfulness.
Smoking status | Baseline, 3, and 12 months.
  Smoking status will be measured as dichotomous outcome (yes or no). If yes, the amount of cigarettes smoked per day will be recorded.
Alcohol use | Baseline, 3, and 12 months.
  Alcohol use will be measured as dichotomous outcome (yes or no). If yes, the number of glasses of alcohol per week will be recorded.
Body Mass Index (BMI) | Baseline, 3, and 12 months.
  BMI will be reported as kg/m².
Blood pressure | Baseline, 3, and 12 months.
  Systolic and diastolic blood pressure will be measured using an automatic monitor. The mean of three measurements will be recorded.
Heart rate | Baseline, 3, and 12 months.
  Heart rate will be measured using an automatic monitor. The mean of three measurements will be recorded.
Serum lipids | Baseline, 3, and 12 months.
  Serum levels of total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides will be reported in units of mmol/L.
Glycated hemoglobin (HbA1c) | Baseline, 3, and 12 months.
  Glycated hemoglobin (HbA1c) will be reported in units of mmol/L.
Cost-effectiveness | 12 months
  The EQ-5D-5L questionnaire will be used for estimating preference weight for health status, which is combined with time in order to compute quality-adjusted life years (QALYs). The cost-effectiveness analysis includes health-care and non-health-care costs and is performed on an intention-to-treat basis. Outcomes are the total costs and QALYs. From these costs and QALYs incremental cost-effectiveness ratios (ICERs) are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Rouwet, MD, PhD, Principal Investigator — Erasmus Medical Center; Joep Teijink, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (2):
- Netherlands (2):
  - Catharina Hospital, Eindhoven
  - Máxima Medical Center, Veldhoven

IPD SHARING:
Plan to Share IPD: No